CLINICAL TRIAL: NCT04456855
Title: Locoregional Surgery of the Primary Tumor in de Novo Stage IV Breast Cancer Patients
Acronym: SYSBTC-001
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-2018-018
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Breast Neoplasm Female; Surgery; Advanced Breast Cancer
Keywords: Breast Neoplasm Female; Locoregional surgery; In de novo stage IV brest cancer; Overall survival; Locoregional progression free survival; Distant progression free survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Locoregional surgery
  Interventions: Procedure: Locoregional surgery
- No surgery

INTERVENTIONS:
Procedure: Locoregional surgery — Patients had pathologically confirmed operable stage IV breast infiltrating carcinoma at initial presentation, and had locoregional surgery for the breast cancer.
  Groups: Locoregional surgery

SUMMARY:
Current guidelines lack definitive evidences about the relative benefits of locoregional surgery for the primary tumor in de novo stage IV breast cancer. The aim of this study (SYSBTC-001) was to investigate the role of locoregional surgery for primary tumor in de novo stage IV breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Operable stage IV breast cancer patients,whose primary lesion is invasive breast cancer confirmed by pathology, and metastases can be confirmed by pathology or imageology examination.
* ECOG-PS 0-2.
* Bone marrow, liver and kidney should be fully functional.
* Patients received the locoregional surgery of the primary tumor in de novo in our center, or didn't received the locoregional surgery of the primary tumor in de novo.
* For the patient who accepted systematic treatment before operation, the systematic treatment must be administered within a year since diagnosed.

Exclusion Criteria:

* Accompanied with other primary malignant tumors.
* Patients who can't plan for follow-up effectively and regularly.
* Multiple liver metastasis and ALT/AST four times higher than normal at patients' first diagnosis.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Operable stage IV breast cancer patients, whose primary lesion is invasive breast cancer confirmed by pathology, and metastases can be confirmed by pathology or imaginology examination
Sampling Method: Non-Probability Sample
Enrollment: 358 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The association between locoregional surgery and overall survival (OS), which defined as the time from the beginning of diagnosis of breast cancer to the death with any causes.

SECONDARY OUTCOMES:
Locoregional progression free survival | 5 years
  Defined as time between the time of diagnosis and the time of locoregional recurrence, or death occurred.
Distant progression free survival | 5 years
  Distant disease free survival (D-DFS), which defined as the time from the diagnosis of de novo stage IV breast cancer to the confirmed time of distant progression, or death due to any other cause.

CONTACTS AND LOCATIONS:
Overall Officials: Herui Yao, PhD, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Jun Tang, PhD, Principal Investigator — Sun Yat-sen University; Guolin Ye, PhD, Principal Investigator — First People's Hospital of Foshan
Locations (3):
- China (3):
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-sen, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu Y, Hong H, Wang Y, Fu T, Chen Y, Zhao J, Chen P, Cai R, Tan Y, He Z, Ren W, Zhou L, Huang J, Tang J, Ye G, Yao H. Clinical Evidence for Locoregional Surgery of the Primary Tumor in Patients with De Novo Stage IV Breast Cancer. Ann Surg Oncol. 2021 Sep;28(9):5059-5070. doi: 10.1245/s10434-021-09650-3. Epub 2021 Feb 3. PMID 33534046